CLINICAL TRIAL: NCT05613426
Title: Effect of Very Early and Rapid Lowering Cholesterol With Evolocumab on Left Ventricular Remodeling in Patients With Anterior ST Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention (EVALUATE-STEMI Trial): a Prospective, Multicenter, Open-label, Adjudicator-blinded, Randomized Clinical Trial
Brief Title: Effect of Very Early and Rapid Lowering Cholesterol With Evolocumab on Left Ventricular Remodeling in Patients With Anterior STEMI Undergoing Primary PCI
Acronym: EVALUATE-STEMI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Principal Investigator, Chuanyu Gao, Vice President, Chief of Cardiology Department, Henan Institute of Cardiovascular Epidemiology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HenanICE202204
Record Dates: First submitted 2022-10-18; First posted 2022-11-14 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: ST Elevation Myocardial Infarction (STEMI)
Keywords: ST Elevation Myocardial Infarction; percutaneous coronary intervention; PCSK9 Inhibitors; left ventricular remodeling
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Ventricular Remodeling | interventions — Rosuvastatin Calcium; evolocumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intensive statin group (Active Comparator): Rosuvastatin, 20 mg per day after randomization
  Interventions: Drug: Rosuvastatin 20 mg
- Combined intensive statin and PCSK9 inhibitor group (Experimental): Evolocumab, 140 mg twice a month after randomization, and Rosuvastatin, 20 mg per day after randomization
  Interventions: Drug: Rosuvastatin 20 mg; Drug: Evolocumab 140 mg/1 ml Subcutaneous Solution [REPATHA]
- PCSK9 inhibitor alone group (Experimental): Evolocumab, 140 mg twice a month after randomization
  Interventions: Drug: Evolocumab 140 mg/1 ml Subcutaneous Solution [REPATHA]

INTERVENTIONS:
Drug: Rosuvastatin 20 mg — Very early use of Rosuvastatin before primary PCI in anterior STEMI
  Arms: Combined intensive statin and PCSK9 inhibitor group; Intensive statin group
Drug: Evolocumab 140 mg/1 ml Subcutaneous Solution [REPATHA] — Very early use of Evolocumab before primary PCI in anterior STEMI
  Arms: Combined intensive statin and PCSK9 inhibitor group; PCSK9 inhibitor alone group

SUMMARY:
For patients with anterior ST elevation myocardial infarction (STEMI) undergoing primary percutaneous coronary intervention (PCI), whether early application of proprotein convertase subtilisin kexin type 9 (PCSK9) inhibitors to rapidly reduce low-density lipoprotein cholesterol (LDL-C) before PCI could effectively inhibit left ventricular remodeling has been rarely reported. The aim of this study was to investigate the effect of early application of PCSK9 inhibitors Evolocumab to rapidly reduce LDL-C levels before primary PCI treatment on left ventricular remodeling in STEMI patients.

Eligible patients were randomly randomized 1:1:1 to one of the following three groups immediately after enrollment: (1) Intensive statin group: rosuvastatin 20 mg per day, in addition to usual therapy; (2) Combined intensive statin and PCSK9 inhibitor group: rosuvastatin 20 mg per day and subcutaneous injection of evolocumab 140 mg twice a month, for at least 3 months, and preferably 6 months; (3) PCSK9 inhibitor alone group: subcutaneous injection of evolocumab 140 mg, twice a month for at least 3 months and preferably 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Persistent chest pain or chest discomfort
* Onset within 12 hours
* ST-segment elevation ≥0.1 millivolt in two adjacent precordial leads, or a new-onset left bundle branch block with dynamic changes
* Primary PCI is planned

Exclusion Criteria:

* Contraindications to Statins or PCSK9 inhibitors
* Prior intravenous thrombolytic therapy
* Prior use of Statins, PCSK9 inhibitors or Ezetimibe
* Cardiogenic shock
* Acute heart failure or pulmonary edema
* Prior chronic heart failure
* Severe hepatic and renal insufficiency (alanine aminotransferase ≥5 upper limit of normal; estimated glomerular filtration rate <30ml/min/1.73m2, or on dialysis)
* Prolonged (> 20 minutes) cardiopulmonary resuscitation
* Definite mechanical complications (including ventricular septal perforation, or rupture of the Papillary tendon bundle, or rupture of the left ventricular free wall)
* Malignant arrhythmias that are difficult to control with drugs
* Severe chronic obstructive pulmonary disease or respiratory failure
* Severe infection
* Neurological disorders
* Bleeding history of cerebrovascular, gastrointestinal, respiratory, urinary or other organs within the last month
* Active bleeding or bleeding diatheses
* Use of anticoagulants
* Malignant tumors or other pathophysiological conditions with an expected survival time of less than 1 year
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in left ventricular ejection fraction (LVEF) | Baseline and 12 weeks
  Echocardiography Core Laboratory, blinded analysis

SECONDARY OUTCOMES:
Change in left ventricular end diastolic/systolic diameter | Baseline and 12 weeks
  Echocardiography Core Laboratory, blinded analysis
Change in left ventricular end diastolic/systolic volume | Baseline and 12 weeks
  Echocardiography Core Laboratory, blinded analysis
A composite of cardiovascular death, recurrent myocardial infarction, ischemic stroke, and hospitalization for heart failure | 12 weeks, 52 weeks
Proportion of LDL-C < 1.4 mmol/L | One week, 12 weeks
Thrombolysis in Myocardial Infarction (TIMI) flow grade | TIMI flow in culprit coronary artery at first coronary angiography, and immediately after primary PCI within 12 hours of onset
Level of troponin | 24 hours, 48 hours, and at hospital discharge, an average of 10 days after randomization
Number of patients with adverse events and serious adverse events | At hospital discharge, an average of 10 days after randomization

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - The People's Hospital of Gongyi, Gongyi, Henan
  - Kaifeng Central Hospital, Kaifeng, Henan
  - The People's Hospital of Changyuan, Xinxiang, Henan
  - Hopeshine Minsheng Hospital of Xinzheng, Xinzheng, Henan
  - The People's Hospital of Xuchang, Xuchang, Henan
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan